CLINICAL TRIAL: NCT06350370
Title: Short-term and Long-term Outcomes of Colorectal Cancer Treated With Natural Orifice Specimen Extraction Surgery : a National Registry-based Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3489
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Natural orifice specimen extraction surgery; Minimally invasive surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NOSES group (Experimental): Patients with colorectal cancer underwent transanal or transvaginal specimen extraction
  Interventions: Procedure: Natural orifice specimen extraction

INTERVENTIONS:
Procedure: Natural orifice specimen extraction — We perform laparoscopic colorectal cancer resection, intracorporeal anastomosis and transanal or transvaginal specimen extraction

SUMMARY:
Natural orifice specimen extraction surgery (NOSES) has gained widespread recognition among scholars and has gradually been promoted and popularized around the world. However, the development of NOSES is still in the exploratory stage and there is a lack of strong evidence from evidence-based medicine to support its feasibility and safety, which has greatly affected its clinical application and development. Based on this, at the call of Professor Xishan Wang, the Chinese NOSES Alliance conducted a large retrospective clinical study involving multiple centers. By summarizing the NOSES cases of nearly 100 centers in China, the study aims to clarify the current status of NOSES surgery in China. Additionally, a comprehensive analysis and summary was conducted by combining the basic information of NOSES patients, perioperative data, postoperative pathological data, and follow-up information to further demonstrate the safety and feasibility of NOSES in the treatment of colorectal cancer. This study also provides more real and objective evidence-based medicine support for the promotion and development of NOSES surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of primary malignant tumor in the colon or rectum;
2. The surgery meets the definition in the "Consensus of NOSES Experts in Colorectal Cancer";

Exclusion Criteria:

1. Postoperative pathological diagnosis does not belong to primary malignant tumors in the colon or rectum;
2. The surgery does not meet the definition in the "Consensus of NOSES Experts in Colorectal Cancer".

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of short-term complication | 30 days after surgery
  Rate of complications occurred within 30 days after surgery

SECONDARY OUTCOMES:
Operative duration | 7 days
  Total time of the operation
Intraoperative blood loss | 7 days
  Estimated blood loss during the surgery
Time to first flatus after surgery | 7 days
  Time to first flatus after surgery
Time to first stool after surgery | 7 days
  Time to first stool after surgery
Length of stay after surgery | 7 days
  Length of stay after surgery
3-year disease free survival | 3 year
  3-year disease free survival
3-year overall survival | 3 year
  3-year overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No